CLINICAL TRIAL: NCT00230672
Title: Studies of Plasma Proteins Derived From Pulmonary Arteriovenous Malformation Patients
Brief Title: Investigation of Plasma Proteins in Patients With Hereditary Haemorrhagic Telangiectasia and PAVMs
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IC/CLS7
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Telangiectasia, Hereditary Hemorrhagic
Keywords: Hereditary Hemorrhagic
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT, also known as Osler-Weber-Rendu Syndrome) is an disease that leads to the development of dilated and fragile blood vessels, including arteriovenous malformations in the lungs (PAVMs). We hypothesize that the genetically-determined abnormality in the blood vessels of HHT patients leads to alteration in the concentrations or activity of several proteins in the blood stream. We propose to take blood samples from patients at defined times in order to study changes in blood protein levels and activity

ELIGIBILITY:
Inclusion Criteria:Patients with hereditary haemorrhagic telangiectasia and pulmonary arteriovenous malformations -

Exclusion Criteria:Unable to provide informed consent

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hereditary haemorrhagic telangiectasia and pulmonary arteriovenous malformations
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2005-03 (Actual); Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Shovlin, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Hammersmith Campus, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Howard LSGE, Santhirapala V, Murphy K, Mukherjee B, Busbridge M, Tighe HC, Jackson JE, Hughes JMB, Shovlin CL. Cardiopulmonary exercise testing demonstrates maintenance of exercise capacity in patients with hypoxemia and pulmonary arteriovenous malformations. Chest. 2014 Sep;146(3):709-718. doi: 10.1378/chest.13-2988. PMID 24676541